CLINICAL TRIAL: NCT03544372
Title: An Investigation Into the Reliability of Self-reported Concussion History in Current Rugby Union Players
Brief Title: Reliability of Self-reported Concussion History in Current Rugby Union Players
Status: Completed | Type: Observational
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Joice Cunningham, Prinicpal Investigator, Ms Joice Cunningham (Phd Candidate), University of Dublin, Trinity College
Other Study IDs: JCunningham2
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Concussion, Mild
Keywords: concussion, rugby, self-report, concussion history, reliability
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Assessment of Concussion History using NIH Concussion History Tool — NIH concussion tool

SUMMARY:
Perhaps no issue in sports medicine has attracted so much media attention and academic interest in recent years as the potential long-term neurodegenerative sequelae of sports-related concussion on athlete's brain health. Rugby has a high incidence of concussion. Recent research findings from a cohort of former professional players found that the number of concussions sustained during their professional careers was associated with the rate of diagnosed clinical depression and late-life cognitive impairment. A limitation of these studies is the use of a self-reported history of concussion. The reliability of professional rugby players to recall and self-report concussion history has never been quantified in the literature to date. Imperfect recall can generate bias in epidemiologic studies when the proportion of events recalled is associated with the health end points of interest. Associations observed may be spurious and due to recall bias if athletes differ in their knowledge and recognition of concussion symptomology in a manner that is associated with the health outcome of interest ie. under/overreporting of concussion. It is difficult to estimate the magnitude of the bias in the absence of any "gold-standard" measure of concussion history. Due to these concerns about the quality of self-reported concussion history, the investigators considered that it was important to evaluate the reliability of self-reported concussion history.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the reliability of self-reported concussion history in current rugby union players

Objectives:

The objectives will be to:

Investigate player's self-report history of sports-related concussion (number and nature of concussions) in this elite rugby playing group.

Correlate player self-report with established individual player medical data. Repeat this process approximately 6 months later on a sub sample of this cohort, in order to test the reliability of player's reported concussion.

ELIGIBILITY:
Inclusion Criteria:

•> 18 years old

* Contracted to Leinster rugby as a professional rugby player
* Players who have given informed consent and are willing to participate in the study.
* Players with a history of sports-related concussion/mild traumatic brain injury.

Exclusion Criteria:

• Any players with a history of non-sports related concussion/severe traumatic brain injury due to road traffic collisions etc. will be excluded.

Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — male
Study Population: current professional rugby union players
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Self-report Concussion History | 30 minutes
  reliability study, agreement between self-report history of concussion via the NIH concussion history tool and documented concussion history. The higher the intraclass correlation between the two-the greater the reliability of the NIH concussion tool

CONTACTS AND LOCATIONS:
Locations (1):
- Trinity College Dublin, Dublin, Ireland